CLINICAL TRIAL: NCT03720197
Title: Registry of Individuals With Type 1 Diabetes Living in Canada: The BETTER Registry
Brief Title: Registry of Patients Living With Type 1 Diabetes
Status: Recruiting | Type: Observational
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Full professor, Institut de Recherches Cliniques de Montreal
Other Study IDs: BETTER
Record Dates: First submitted 2018-10-19; First posted 2018-10-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Waist Circumference; Blood Specimen Collection; Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants aged less than 14 years old
  Interventions: Other: Online questionnaire - Phase 1; Other: Continuous glucose monitor
- Participants aged 14 years old and older
  Interventions: Other: Online questionnaire - Phase 1; Other: Online questionnaire - Phase 2; Other: Online questionnaire - Phase 3; Other: Food questionnaire; Other: Pedometer; Other: Waist circumference; Other: Blood and urine tests; Other: List of medications; Other: Continuous glucose monitor

INTERVENTIONS:
Other: Online questionnaire - Phase 1 — Draw an overall picture of the population with type 1 diabetes in Canada in terms of demographics, diabetes treatment, hypoglycemia frequency and diabetes complications.
Other: Online questionnaire - Phase 2 — Characterize the causes, experience and consequences of hypoglycemia.
  Groups: Participants aged 14 years old and older
Other: Online questionnaire - Phase 3 — Collect information on diabetes and hypoglycemia treatment, hyperglycemia management, sleep habits, depression, physical activity and the benefits of technologies to reduce the frequency of hypoglycemia.
  Groups: Participants aged 14 years old and older
Other: Food questionnaire — 24-hour food recall questionnaire
  Groups: Participants aged 14 years old and older
Other: Pedometer — Participants will wear a podometer for 14 consecutives days
  Groups: Participants aged 14 years old and older
Other: Waist circumference — Participants will be asked to measure their waist circumference
  Groups: Participants aged 14 years old and older
Other: Blood and urine tests — Participants will be invited to send us their latests blood and urine test results.
  Groups: Participants aged 14 years old and older
Other: List of medications — Participants will be invited to send us their list of medications
  Groups: Participants aged 14 years old and older
Other: Continuous glucose monitor — Participants will be invited to send us the latest report of their continuous glucose monitor

SUMMARY:
A registry of individuals with type 1 diabetes open to all patients with type 1 diabetes living in Canada will be established. The objective of this registry will be to measure the frequency and the severity of episodes of hypoglycemia. Participants will be invited to answer questionnaires about the frequency of their hypoglycemic episodes, their fear about hypoglycemia, their symptoms of hypoglycemia, the factors in cause (insulin therapy, nutrition, exercise, etc.), etc.

Participation to the registry is divided in 3 phases. The first phase is mandatory for all participants. Phases 2 and 3 are optional.

DETAILED DESCRIPTION:
The objective of phase 1 is to draw an overall picture of the population with type 1 diabetes in Canada in terms of demographics, diabetes treatment, hypoglycemia frequency and diabetes complications. It takes about 10 minutes to answer the questionnaire. If the participant uses a continuous glucose monitor and agrees, the participant is invited to send the latest report of the continuous glucose monitor.

The objective of phase 2 is to characterize the causes, experience and consequences of hypoglycemia. Phase 2 also involves, if the participant accepts and live in the province of Quebec or Alberta, to provide the research team with their latest blood and urine tests as well as their list of medications.

The objective of phase 3 is to collect information on diabetes and hypoglycemia treatment, hyperglycemia management, sleep habits, depression, physical activity and the benefits of technologies to reduce the frequency of hypoglycemia. Phase 3 also involves, if the participant agrees, answering a food questionnaire, wearing a step counter, measuring waist circumference

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes
* Living in Canada

Exclusion Criteria:

* Type 2 diabetes
* Gestational diabetes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with type 1 diabetes living in Canada.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of non-severe hypoglycemic episodes | 12 months
  Participants will be asked to report the number of non-severe hypoglycemic episodes in the last 12 months in a questionnaire designed by the investigators. The definition of non-severe hypoglycemia is a blood sugar below 3.0 mmol/L that the participant was able to treat himself

SECONDARY OUTCOMES:
Number of severe hypoglycemic episodes | 12 months
  Participants will be asked to report the number of severe hypoglycemic episodes in the last 12 months in a questionnaire designed by the investigators. The definition of severe hypoglycemia is low blood sugar levels requiring help from another person or use of glucagon or hospitalization or loss of consciousness.
Fear of hypoglycemia | 6 months
  Fear of hypoglycemia will be assessed by the Hypoglycemia Fear Survey II.
Diabetes distress | 1 month
  Diabetes distress will be assessed by the Diabetes Distress Scale.
Medical follow-up for diabetes | 12 months
  Participants will be asked to report in a questionnaire designed by the investigators how many times in the last 12 months they have seen a health care professionals (family doctor, medical specialist, nurse, nutritionnist, kinesiologist, psychologist, pharmacist, social worker).
Insulin doses | 3 days
  Participants will be asked to report in a questionnaire designed by the investigators their insulin doses of the last 3 days (basal insulin and insulin given at mealtime).
Physical activity | 1 week
  Physical activity will be assessed by the International Physical Activity Questionnaire.
Sleep habits | 1 month
  Sleep habits will be assessed by the Pittsburgh Sleep Quality Index
Depression | 2 weeks
  Depression will be assessed by the Patient Health Questionnaire (PHQ-9)
Number of steps | 14 days
  The number of steps will be measured by a pedometer

CONTACTS AND LOCATIONS:
Overall Officials: Remi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (7):
- Canada (7):
  - Alberta Diabetes Institute, Edmonton, Alberta
  - Institut de recherches cliniques de Montréal, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Centre Hospitalier Universitaire de Québec-Université Laval, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Housni A, Katz A, Kichler JC, Nakhla M, Secours L, Brazeau AS. Predictors of stigma perception by people with type 1 diabetes: A cross-sectional analysis of the BETTER registry. Diabetes Metab Syndr. 2024 Aug;18(8):103112. doi: 10.1016/j.dsx.2024.103112. Epub 2024 Aug 29. PMID 39236506
- [Background] Lalanne-Mistrih ML, Bonhoure A, Messier V, Boudreau V, Lebbar M, Talbo MK, Sun CJ, Bandini A, Secours L, Calderon V, Grou C, Tressieres B, Brazeau AS, Rabasa-Lhoret R. Overweight and Obesity in People Living With Type 1 Diabetes: A Cross-Sectional Analysis of the BETTER Registry. Diabetes Metab Res Rev. 2024 Sep;40(6):e3837. doi: 10.1002/dmrr.3837. PMID 39193662
- [Background] Madar H, Lalanne-Mistrih ML, Lebbar M, Wu Z, Robitaille Y, Pelletier J, Grou C, Brazeau AS, Rabasa-Lhoret R. Cardiovascular Risk Factors and Adherence to Cardiovascular Protection Practice Guidelines in Adults With Type 1 Diabetes: A BETTER Registry Cross-sectional Analysis. Can J Diabetes. 2023 Aug;47(6):473-481.e1. doi: 10.1016/j.jcjd.2023.04.006. Epub 2023 Apr 12. PMID 37059389
- [Background] Wu Z, Talbo M, Lebbar M, Messier V, Courchesne A, Brazeau AS, Rabasa-Lhoret R. Characteristics associated with having a hemoglobin A1c </= 7 % (</=53 mmol/mol) among adults with type 1 diabetes using an automated insulin delivery system. Diabetes Res Clin Pract. 2023 Dec;206:111006. doi: 10.1016/j.diabres.2023.111006. Epub 2023 Nov 10. PMID 37952601
- [Background] Talbo MK, Lebbar M, Wu Z, Vanasse A, Lalanne-Mistrih ML, Brazeau AS, Rabasa-Lhoret R. Gender differences in reported frequency and consequences of hypoglycemia among adults living with type 1 diabetes: Results from the BETTER registry. Diabetes Res Clin Pract. 2023 Aug;202:110822. doi: 10.1016/j.diabres.2023.110822. Epub 2023 Jul 7. PMID 37423499
- [Background] Wu Z, Rabasa-Lhoret R, Messier V, Shohoudi A, Dasgupta K, Pelletier J, Brazeau AS. Self-reported haemoglobin A1c highly agrees with laboratory-measured haemoglobin A1c among adults living with type 1 diabetes: A BETTER registry study. Diabetes Metab. 2022 Jan;48(1):101277. doi: 10.1016/j.diabet.2021.101277. Epub 2021 Sep 9. No abstract available. PMID 34509633
- [Background] Nguyen E, Wong K, Lalanne-Mistrih ML, Rabasa-Lhoret R, Brazeau AS. Association between low-carbohydrate-diet score, glycemia and cardiovascular risk factors in adults with type 1 diabetes. Nutr Metab Cardiovasc Dis. 2024 Sep;34(9):2143-2154. doi: 10.1016/j.numecd.2024.04.014. Epub 2024 Apr 27. PMID 38866607
- [Background] Talbo MK, Katz A, Dostie M, Legault L, Brazeau AS. Associations Between Socioeconomic Status and Patient Experience With Type 1 Diabetes Management and Complications: Cross-sectional Analysis of a Cohort From Quebec, Canada. Can J Diabetes. 2022 Aug;46(6):569-577. doi: 10.1016/j.jcjd.2022.02.008. Epub 2022 Mar 3. PMID 35864032
- [Background] Talbo MK, Rabasa-Lhoret R, Yale JF, Peters TM, Brazeau AS. Are nocturnal hypoglycemia prevention strategies influenced by diabetes technology usage? A BETTER registry analysis. Diabetes Res Clin Pract. 2022 Sep;191:110080. doi: 10.1016/j.diabres.2022.110080. Epub 2022 Sep 12. PMID 36099973
- [Background] Prevost MS, Rabasa-Lhoret R, Talbo MK, Yardley JE, Curry EG, Brazeau AS. Gender Differences in Strategies to Prevent Physical Activity-Related Hypoglycemia in Patients With Type 1 Diabetes: A BETTER Study. Diabetes Care. 2022 Mar 1;45(3):e51-e53. doi: 10.2337/dc21-1899. No abstract available. PMID 35045175
- [Derived] Madar H, Wu Z, Bandini A, Perkins B, Messier V, Pomey MP, Brazeau AS, Rabasa-Lhoret R. Influence of severe hypoglycemia definition wording on reported prevalence in adults and adolescents with type 1 diabetes: a cross-sectional analysis from the BETTER patient-engagement registry analysis. Acta Diabetol. 2023 Jan;60(1):93-100. doi: 10.1007/s00592-022-01987-9. Epub 2022 Oct 17. PMID 36245008
- [Derived] Brazeau AS, Messier V, Talbo MK, Gagnon C, Taleb N, Fortier I, Wu Z, Perkins BA, Carpentier AC, Bandini A, Rabasa-Lhoret R; BETTER Study Group. Self-reported Severe and Nonsevere Hypoglycemia in Type 1 Diabetes: Population Surveillance Through the BETTER Patient Engagement Registry: Development and Baseline Characteristics. Can J Diabetes. 2022 Dec;46(8):813-821. doi: 10.1016/j.jcjd.2022.05.010. Epub 2022 May 28. PMID 35835670